CLINICAL TRIAL: NCT01090986
Title: Prediction of Home Mechanical Ventilation Effectiveness by Means of Non-controlled Air Leaks Estimation.
Brief Title: Home Mechanical Ventilation Effectiveness and Air Leaks
Status: Completed | Type: Observational
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: PR02/02/2007
Record Dates: First submitted 2010-03-19; First posted 2010-03-23 (Estimated); Last update posted 2014-02-24 (Estimated); Status verified 2014-02

CONDITIONS: Pulmonary Disease; Chronic Respiratory Failure; COPD
Keywords: Restrictive pulmonary disease with hypercapnic chronic respiratory failure.; COPD patients who need NIV hypercapnic chronic respiratory failure.
MeSH Terms: conditions — Lung Diseases; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients with a restrictive pulmonary disease and hypercapnic chronic respiratory failure with standard criteria for NIV. Also COPD patients who need NIV because of another reason (obesity, nocturnal hyperventilation or nocturnal hypercapnic response to oxygen).

SUMMARY:
Non invasive ventilation (NIV) usually presents air leaks that may determine the result of this treatment. The clinical usefulness of analyzing (and quantifying) these leaks during the adaptation period to NIV has not been evaluated in prospective clinical studies as a predictive data of treatment effectiveness. Our hypothesis is that air leaks are correlated to a successful adaptation to NIV. And air leak magnitude may predict early failures of this treatment. And also, as we do not know if air leaks change during the adaptation period to NIV, we do not know whether early detection of air leaks plays a role in the therapeutic outcome. Our objective is to evaluate the clinical usefulness of quantifying air leaks during the adaptation period to NIV as a predictor of effectiveness of this treatment. We also want to evaluate the correlation between air leaks and clinical-functional patients' profile, and the ventilatory parameters selected and to evaluate air leaks variability during the adaptation period to NIV. Method: We will determine the air leak magnitude in twenty patients during adaptation to NIV. We will use VPAP III ventilators (ResMed, Australia), commercial nasal masks (Mirage o Ultra Mirage) and VPAP III/ResLinkTM (ResMed, North Ryde, Australia), a device that includes a monitoring system coupled with the VPAP III ventilator. This device allows to record air leaks and other ventilation parameters. We will perform four VPAP III/ResLinkTM recordings in each patient (the last night in hospital during the adaptation period, the first night at home, and one and two months later, after the initiation of NIV treatment). We will also perform a complete pulmonary function test, quality-of-life questionnaire (SF36), and a tolerance to NIV questionnaire in all patients at the onset of NIV treatment and two months later. We will evaluate which patients will need to change treatment at the end of the adaptation period to NIV. We also will analyze and compare air leaks magnitude in each of the four recordings stated above.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a restrictive pulmonary disease (slow evolution neuromuscular or thorax cage diseases, obesity or nocturnal hypoventilation) and hypercapnic chronic respiratory failure with standard criteria for NIV.
* COPD patients who need NIV because of another reason (obesity, nocturnal hyperventilation or nocturnal hypercapnic response to oxygen).
* PaCO2 ≥ de 50 mmHg.
* Clinically stable (at least for one month).
* Possibility to fit a nasal mask for NIV treatment (ultra mirage, mirage).

Exclusion Criteria:

* Rapid evolution neuromuscular disease (Amyotrophic Lateral Sclerosis).
* Serious comorbidity.
* Lack of patients comprehension or collaboration.
* Inability to fit a nasal mask for NIV treatment (ultra mirage, mirage).
* Treatment compliance < 4h/d.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: * Patients with a restrictive pulmonary disease (slow evolution neuromuscular or thorax cage diseases, obesity or nocturnal hypoventilation) and hypercapnic chronic respiratory failure with standard criteria for NIV.
  * Also COPD patients who need NIV because of another reason (obesity, nocturnal hyperventilation or nocturnal hypercapnic response to oxygen).
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2006-06; Primary Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Clinical usefulness of quantifying AIR LEAKS during the adaptation period to NIV as a predictor of effectiveness (pCO2 EVOLUTION) of this treatment. | One year

SECONDARY OUTCOMES:
- Air leaks AND patients' characteristics.- Some indices (air leaks/inspiratory pressure...)and NIV effectiveness. - Air leak evolution.- Air leaks and patients' tolerance to NIV. | One year

CONTACTS AND LOCATIONS:
Overall Officials: Carme Puy, MD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona, Spain